CLINICAL TRIAL: NCT03492060
Title: Neurogenetic Disorders: A Longitudinal Study on Natural History and Intervention Strategies
Brief Title: Longitudinal Study of Neurogenetic Disorders
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Simons Foundation (Other); New York University (Other); Hackensack Meridian Health (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: AAAR7203
Record Dates: First submitted 2018-04-02; First posted 2018-04-10 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Neurodevelopmental Disorders; Intellectual Disability; Developmental Delay; Autism Spectrum Disorder; Seizures; Hypertonia, Muscle; Hypotonia
Keywords: Gene Variant; HNRNPA1; HNRNPA2; HNRNPB1; HNRNPC1; HNRNPC2; HNRNPD; HNRNPE1; HNRNPE2; HNRNPE3; HNRNPE4; HNRNPG; HNRNPH1; HNRNPH2; HNRNPI; HNRNPK; HNRNPL; HNRNPM; HNRNPP; HNRNPQ1; HNRNPQ2; HNRNPQ3; HNRNPR; HNRNPU
MeSH Terms: conditions — Neurodevelopmental Disorders; Intellectual Disability; Learning Disabilities; Autism Spectrum Disorder; Seizures; Muscle Hypertonia; Muscle Hypotonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood and tissue samples will be obtained through one of three ways:
  1. The sample can be taken as part of routine clinical care; for example, by a referring physician, and sent to our site for storage.
  2. An existing sample you may have provided for research in another study can be transferred to our site for storage.
  3. The sample can be taken by the Principal Investigator of this study for research and will be stored at our site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Variant in a hnRNP gene: Individuals with a variant in any hnRNP gene who present with neurodevelopmental abnormalities are eligible for the study.
- Variant in other gene: Individuals with a confirmed variant in other genes who present with neurodevelopmental abnormalities are eligible for the study.

SUMMARY:
The purpose of this study is to analyze patterns in individuals with hnRNP (and other) genetic variants, including their neurological comorbidities, other medical problems and any treatment. The investigators will maintain an ongoing database of medical data that is otherwise being collected for routine medical care. The investigators will also collect data prospectively in the form of questionnaires, neuropsychological assessments, motor assessments, and electroencephalography to examine the landscape of deleterious variants in these genes.

DETAILED DESCRIPTION:
Neurodevelopmental disorders are a group of disorders in which the development of the central nervous system is disturbed. The genetic basis for many neurodevelopmental disorders has continued to expand and a recent gene called HNRNPH2 (Heterogeneous Nuclear Ribonucleoprotein H2, encoded by HNRNPH2) is one such gene that is associated with a common neurodevelopmental disorder characterized by developmental delay, intellectual disability, autism and autistic features, and tone abnormalities, among other multisystem problems.

The investigators will expand the genetic cohort to include any individual with a confirmed variant in any gene presenting with neurodevelopmental abnormalities. This is non-interventional study that examines both data previously used in clinical practice and prospective data collection in the form of questionnaires and assessments. The investigators will examine patterns of initial presentation, patterns in neurological evaluations; neurological testing including brain MRI and electroencephalography, and outcomes in individuals with genetic variants.

Genes of Focus:

hnRNPA1 hnRNPA2 hnRNPB1 hnRNPB2 hnRNPC2 hnRNPD hnRNPE1 hnRNPE2 hnRNPE3 hnRNPE4 hnRNPG hnRNPH1 hnRNP H2 hnRNPI hnRNPK hnRNPL hnRNPM hnRNPP hnRNPQ1 hnRNPQ2 hnRNPQ3 hnRNPR hnRNPU

ELIGIBILITY:
Inclusion Criteria:

* Individuals must have had whole genome/exome sequencing and have a confirmed variant in any gene.

Exclusion Criteria:

* Subjects who cannot provide genetic confirmation of a predicted deleterious variant in any gene.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have already undergone genetic testing and carry a variant in any gene. Individuals will often present with neurological abnormalities, although the absence of symptoms is not exclusion criterion for the study. International subjects are welcome to enroll if eligibility criteria is met.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Medical abnormalities associated with genetic variants | 5 years
  Gene variants are known to result in a variety of clinical phenotypes. The study is intended to accrue data from medical records that document the range of neurological phenotypes and explore their incidence and frequency across genetic cohorts.
Education-based impairments associated with genetic variants | 5 years
  The study seeks to collect records from the schools attended by participants; including: Individualized Education Programs (IEPs) and school records. We intend to use these records, in tandem with medical records, to explore meaningful statistical and clinical relationships in the phenotypes expressed by the population of the study.
Repetitive Behavior | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and repetitive behavior (measured by the Repetitive Behavior Scale - Revised; RBS-R)
Sleep Habits | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and sleep habits (measured by The Children's Sleep Habits Questionnaire; CSHQ)
Sensory Issues | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and sensory issues (measured by The Short Sensory Profile; SSP)
Social Interaction and Communication SRS-II Score | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and social interaction and communication issues (measured by The Social Responsiveness Scale - Second Edition; SRS-II)
Anxiety | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and anxiety (measured by The Spence Children's Anxiety Scale - Preschool and Parent Reports; SCAS - Preschool and SCAS - P)
Receptive Language Skills | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and receptive language skills (measured by a 20-item music exposure questionnaire evaluating exposure on a 3-point scale: rarely, sometimes, often; and an EEG with music paradigm)
Executive Functioning | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and executive functioning (measured by The Behavior Rating Inventory of Executive Function - Parent Report; BRIEF-P)
Autism | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and autism (measured by The Childhood Autism Rating Scale; CARS)
Adaptive Behavior | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and adaptive behavior (measured by The Vineland Adaptive Behavior Scales, Third Edition; Vineland - 3)
Social Interaction and Communication SCQ Score | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and social interaction and communication issues (measured by The Social Communication Questionnaire; SCQ)
Emotional Regulation | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and emotional regulation (measured by The Behavioral Assessment System for Children - Third Edition; BASC - 3)
Motor Performance | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and motor performance (measured by The Movement Assessment Battery for Children - Second Edition; MASC-II)
Function in Daily Activities, Mobility, Social and Cognitive, and Responsibility | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and functional capability in daily activities and mobility (measured by The Pediatric Evaluation of Disability Inventory Computer Adaptive Test; PEDI-CAT)
Functional Balance | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and functional balance and gross motor function (measured by a 14-item Pediatric Balance Scale)
Functional Capability and Mobility | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and functional mobility (measured by an 11-point Movement Questionnaire)
Coordination and Gait | 5 years
  Correlations (r) between mutant allele (obtained from retrospective data) and gait (measured by a Kinematic Evaluation utilizing Solesound Pedishoe Sandals and GaitRite Walkway)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M. Bain, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared with the Simons Foundation. This is applicable only to participants dually enrolled in both studies (as stipulated in the consent process). Individual data for all primary and secondary outcome measures will be made available. Subject data will also be shared with affiliated institutions for relevant genotypes, as outlined in the consent process.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available per request as it is accrued throughout the course of the study.
Access Criteria: Data access requests will be reviewed by the PI and study team. Requestors will be required to sign a data access agreement.
URL: https://simonsfoundation.org

REFERENCES:
- [Background] Bain JM, Cho MT, Telegrafi A, Wilson A, Brooks S, Botti C, Gowans G, Autullo LA, Krishnamurthy V, Willing MC, Toler TL, Ben-Zev B, Elpeleg O, Shen Y, Retterer K, Monaghan KG, Chung WK. Variants in HNRNPH2 on the X Chromosome Are Associated with a Neurodevelopmental Disorder in Females. Am J Hum Genet. 2016 Sep 1;99(3):728-734. doi: 10.1016/j.ajhg.2016.06.028. Epub 2016 Aug 18. PMID 27545675
- [Result] Bain JM, Thornburg O, Pan C, Rome-Martin D, Boyle L, Fan X, Devinsky O, Frye R, Hamp S, Keator CG, LaMarca NM, Maddocks ABR, Madruga-Garrido M, Niederhoffer KY, Novara F, Peron A, Poole-Di Salvo E, Salazar R, Skinner SA, Soares G, Goldman S, Chung WK. Detailed Clinical and Psychological Phenotype of the X-linked HNRNPH2-Related Neurodevelopmental Disorder. Neurol Genet. 2021 Jan 29;7(1):e551. doi: 10.1212/NXG.0000000000000551. eCollection 2021 Feb. PMID 33728377
- [Derived] Davis TJ, Salazar R, Beenders S, Boehme A, LaMarca NM, Bain JM. A Prospective, Longitudinal Study of Caregiver-Reported Adaptive Skills and Function of Individuals with HNRNPH2-related Neurodevelopmental Disorder. Adv Neurodev Disord. 2024;8(3):445-456. doi: 10.1007/s41252-023-00346-1. Epub 2023 Aug 7. PMID 39220267
- See also: Original HNRNPH2 genetic cohort website — http://hnrnph2.com